CLINICAL TRIAL: NCT06658392
Title: Domain-general and Domain-specific Contributions to the Development of Numerical Cognition
Acronym: CFDDCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D20-P011
Record Dates: First submitted 2024-10-03; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: No Condition
Keywords: cognitive neuroscience; numerical cognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arithmetic (Experimental): exploring neurocognitive mechanisms underlying development of arithmetic competencies in healthy children.
  Interventions: Other: cognitive tasks

INTERVENTIONS:
Other: cognitive tasks — no intervention in a medical sense, only observing changes of BOLD signal during different experimental conditions in cognitive tasks (arithmetic, attention, inhibition)

SUMMARY:
Exploring the non-symbolic and symbolic arithmetic competencies in two groups of children (5-, and 7-year-olds). Additionally, we explored the relationship with domain-general factors such as inhibition and attention. Recorded fMRI.

DETAILED DESCRIPTION:
Using T2*-weighted eip imaging, we measured BOLD response in two cohorts of healthy children while they were doing different cognitive tasks in the scanner. These tasks included solving non-symbolic (i.e. sets of elements) and symbolic (i.e. Arabic digits) addition and subtraction problems, a color control task, an attentional task measuring different facets of spatial attention, and a task measuring inhibition. We also recorded a high-resolution anatomical scan of the brain.

ELIGIBILITY:
Inclusion Criteria:

* school enrollment
* French as mother tongue
* right-handed
* normal medical, neurological and neuroradiological examinations - parents affiliated to a social security scheme

Exclusion Criteria:

* not within age range
* monocygotic twins
* - contraindications to an MRI examination (neurosensory stimulator or implantable defibrillator, cochlear implants, ferromagnetic ocular or cerebral foreign bodies close to nerve structures, metal prostheses, patient agitation: uncooperative or agitated patients, claustrophobic subjects, ventriculoperitoneal neurosurgical shunt valves, dental apparatus, etc.).
* sudden onset of cognitive problems that could indicate a stroke; a history of head trauma with loss of consciousness lasting more than 1 hour, or encephalitis; - a chronic neurological, psychiatric, endocrine, hepatic or infectious condition
* a history of major illness (diabetes, chronic lung disease, severe cardiac, metabolic, hematological, endocrinological or immunological disorders, cancer); - medication likely to interfere with brain imaging measurements
* color blindness or uncorrected visual disorders
* inability to take part in the study for geographical or psychiatric reasons
* presence of pervasive developmental and/or acquisition disorders identified by parents or legal guardians and/or teachers
* cerebral palsy
* impaired fine motor skills
* parents or legal guardians not affiliated to a social security scheme
* unaccompanied by parent(s) or legal guardian(s) during visits.
* tattoo not compatible with MRI
* children and parents under legal protection

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
BOLD response | BOLD response recorded during fMRI session
  changes of BOLD response under different experimental conditions (non-symbolic arithmetic; symbolic arithmetic; inhibition; attention)
BOLD response | during fMRI session
  changes of BOLD response in experimental conditions

CONTACTS AND LOCATIONS:
Overall Officials: Catherine OPPENHEIM, Pr, Principal Investigator — Promotor
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France